CLINICAL TRIAL: NCT02636582
Title: VADIS Trial: Phase II Trial of Nelipeimut-S Peptide Vaccine in Women With DCIS of the Breast
Brief Title: Nelipepimut-S Plus GM-CSF Vaccine Therapy in Treating Patients With Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: NCI-2015-02189; NCI-2015-02189 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); N01-CN-2012-00034; 2016-0164 (Other: M D Anderson Cancer Center); MDA2014-04-02 (Other: DCP); N01CN00034 (NIH); P30CA016672 (NIH)
Record Dates: First submitted 2015-12-18; First posted 2015-12-22 (Estimated); Results first posted 2023-05-16 (Actual); Last update posted 2023-12-05 (Actual); Status verified 2023-11

CONDITIONS: Breast Ductal Carcinoma In Situ
MeSH Terms: conditions — Carcinoma, Intraductal, Noninfiltrating | interventions — HER2 peptide (369-377); Granulocyte-Macrophage Colony-Stimulating Factor; sargramostim; Colony-Stimulating Factors; Surgical Procedures, Operative

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (nelipepimut-S plus GM-CSF vaccine) (Experimental): Patients receive nelipepimut-S plus GM-CSF vaccine ID on days 0 and 14 and then undergo surgery on day 28.
  Interventions: Other: Laboratory Biomarker Analysis; Drug: Nelipepimut-S Plus GM-CSF Vaccine; Procedure: Surgical Procedure
- Arm II (sargramostim) (Active Comparator): Patients receive sargramostim ID on days 0 and 14 and then undergo surgery on day 28.
  Interventions: Other: Laboratory Biomarker Analysis; Biological: Sargramostim; Procedure: Surgical Procedure

INTERVENTIONS:
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Nelipepimut-S Plus GM-CSF Vaccine — Given ID
  Other Names: E75 Plus GM-CSF; E75 Vaccine Plus GM-CSF; HLA A2/A3-Restricted HER-2/neu Peptide Vaccine Plus GM-CSF; Nelipepimut-S Plus Sargramostim; NeuVax Plus GM-CSF
  Arms: Arm I (nelipepimut-S plus GM-CSF vaccine)
Biological: Sargramostim — Given ID
  Other Names: 23-L-Leucinecolony-Stimulating Factor 2; DRG-0012; Leukine; Prokine; rhu GM-CFS; Sagramostim; Sargramostatin
  Arms: Arm II (sargramostim)
Procedure: Surgical Procedure — Undergo surgery
  Other Names: Operation; Surgery; Surgery Type; Surgery, NOS; Surgical; Surgical Intervention; Surgical Interventions; Surgical Procedures; Type of Surgery

SUMMARY:
This phase II trial studies how well nelipepimut-S plus GM-CSF vaccine therapy or sargramostim works in treating patients with breast cancer. Vaccines made from peptide or antigen and/or a person's white blood cells mixed with tumor proteins may help the body build an effective immune response to kill tumor cells that express breast cancer antigens. It is not yet known whether nelipepimut-S plus GM-CSF vaccine or sargramostim is more effective in treating patients with breast cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Evaluate for nelipepimut-S-specific cytotoxic T lymphocyte (CTL; cluster of differentiation [CD]8+ T cell) response in patients receiving NeuVax (nelipepimut-S plus GM-CSF [sargramostim]) compared to patients receiving GM-CSF alone (control).

SECONDARY OBJECTIVES:

I. Toxicity profile and frequency of adverse events in women with ductal carcinoma in situ (DCIS) of the breast receiving nelipepimut-S vaccine as compared to women receiving GM-CSF alone.

II. Presence of DCIS at resection. III. Difference in HER2 expression in the biopsy and the surgical specimen excised post-vaccination.

IV. Histologic responses:

IVa. Degree of lymphocyte infiltration determined on hematoxylin and eosin (H&E) stained slides and immune infiltration as determined by multiplex immunofluorescence staining for markers including but not limited to CD3, CD4 and CD8.

IVb. Immune infiltrates in normal tissue maximally distant from the tumor (in mastectomy samples).

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I: Patients receive nelipepimut-S plus GM-CSF vaccine intradermally (ID) on days 0 and 14 and then undergo surgery on day 28.

ARM II: Patients receive sargramostim ID on days 0 and 14 and then undergo surgery on day 28.

After completion of study treatment, patients are followed up at 1 and 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be pre- or post-menopausal
* Participants must have a diagnosis of DCIS made by core needle biopsy
* Participants must be human leukocyte antigen (HLA)-A2 positive
* Eastern Cooperative Oncology Group (ECOG) performance status must be 0 or 1 (Karnofsky >= 60%)
* Clinical chemistry less than 2 x normal upper limit of normal range
* Platelets >= 100,000/mm^3
* Hemoglobin >= 10 g/dL
* Blood urea nitrogen < 2 x upper limit of normal (ULN)
* Alkaline phosphatase < 2 x ULN
* Lactate dehydrogenase < 2 x ULN
* Creatinine < 2 x ULN
* Bilirubin < 2 x ULN
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) < 2 x ULN
* A normal ejection fraction, as defined by the participant's institution; only limited echocardiograms (ECHOs) will be used as cardiac evaluation; no other tests are allowed; ECHO is to be done only in HLA-A2 positive participants; if ECHO has been done within 30 days prior to randomization and results showing a normal ejection fraction have been obtained prior to randomization, an additional ECHO is not needed at baseline
* Willingness to comply with all study interventions and follow-up procedures
* The ability to understand and willingness to sign a written informed consent document

Exclusion Criteria:

* Invasive breast cancer; areas of microinvasion or suspicious for microinvasion on the core biopsy is allowed
* History of prior breast cancer treated within the past two years; patients completing all breast cancer-specific treatment over two years prior to the current diagnosis are eligible
* History of prior ductal carcinoma in situ (DCIS) treated within the past two years; patients completing all treatment for a previous diagnosis of DCIS over two years prior to the current diagnosis are eligible
* Prior lobular carcinoma in situ (LCIS) is allowed
* Pregnant, unwilling to use adequate contraception during study treatment duration or breastfeeding; the effects of NeuVax on the developing human fetus are unknown; for this reason and because NeuVax may be teratogenic, pregnant women will be excluded; all heterosexually active women who may become pregnant must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation OR be post-menopausal defined as any one of the following 1) prior hysterectomy, 2) absence of menstrual period for 1 year in the absence of prior chemotherapy or 3) absence of menstrual period for 2 years in women with a prior history of chemotherapy exposure who were pre-menopausal prior to chemotherapy; should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her study physician immediately
* Any autoimmune disease or other medical condition that, in the opinion of the investigator, would compromise the subject's safety
* Immune deficiency diseases such as immunoglobulin deficiency or immunosuppressive therapy that might interfere with appropriate immune response
* Known history of or known active infection with human immunodeficiency virus (HIV), hepatitis B or hepatitis C
* Patients on chronic steroid therapy or other immunosuppressive therapy except for topical or inhaled steroids known to have low systemic absorption
* Patients with a known hypersensitivity to GM-CSF, yeast-derived products, or any component of the GM-CSF product (e.g., mannitol)
* Concurrent treatment with other investigational agent
* History of non-breast malignancy within 5 years prior to randomization, except curatively treated superficial bladder cancer, carcinoma in situ of the cervix (stage 0-1), and basal cell or squamous cell carcinoma of the skin
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to NeuVax
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* No recent or planned immunotherapy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2016-06-14 (Actual); Primary Completion 2019-07-22 (Actual); Study Completion 2023-05-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Powel H Brown, Principal Investigator — M.D. Anderson Cancer Center
Locations (4):
- United States (4):
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - NYP/Columbia University Medical Center/Herbert Irving Comprehensive Cancer Center, New York, New York
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - M D Anderson Cancer Center, Houston, Texas

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Females >/= 18 years with DCIS identified on core needle biopsy and at least 1cm area of radiographic abnormality.
Pre-assignment Details: Only patients with allele HLA-A2 eligible for randomization. 23-were HLA-A2 negative, 7 were HLA-A2 positive and of the 7: 4-withdrew once they received their results, 1- had disease progression, 1-opted for earlier surgery and 1- opted for earlier surgery when trial went on hold after consent.
Groups:
- GM-CSF (Control): Immunoadjuvant GM-CSF
- Nelipepimut-S (NPS+GM-CSF): Vaccine with immunogenic peptide nelipepimut-S+GM-CSF (NPS+GM-CSF)
Period: Overall Study
Arm/Group | GM-CSF (Control) | Nelipepimut-S (NPS+GM-CSF)
Started | 4 | 9
At Surgery | 4 | 9
1- Month Post-Op | 4 | 9
3-6 Months Post-Op | 3 | 9
Completed | 3 | 9
Not Completed | 1 | 0
Not completed — Surgical Pathology | 1 | 0

BASELINE CHARACTERISTICS:
Population: Randomized participants.
Groups:
- Arm I GM-CSF: Immunoadjuvant GM-CSF
- Arm II NPS+GM-CSF: Vaccine with immunogenic peptide nelipepimut-S+GM-CSF (NPS+GM-CSF)
- Total: Total of all reporting groups
Arm/Group | Arm I GM-CSF | Arm II NPS+GM-CSF | Total
Number analyzed (Participants) | 4 | 9 | 13
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 54.5 [43.3 to 65] | 57 [49 to 65] | 57 [47 to 63]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 9 | 13
  Male | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 4 | 9 | 13

OUTCOME MEASURES:

1. Primary Outcome: Mean Percent of Nelipepimut-S-specific Cytotoxic T Lymphocyte Response (E75)
Description: Change from baseline in the Mean percent of Nelipepimut-S-specific cytotoxic T lymphocyte response one-month post-surgical resection. Wilcoxon rank sum test exact P-value was used.
Time Frame: One-Month post-surgical resection from baseline
Measure: Mean (Inter-Quartile Range); unit: percent of cytotoxic T lymphocytes
Groups:
- GM-CSF: Immunoadjuvant GM-CSF
- NPS+GM-CSF: Vaccine with immunogenic peptide nelipepimut-S+GM-CSF (NPS+GM-CSF)
Arm/Group | GM-CSF | NPS+GM-CSF
Number analyzed (Participants) | 4 | 9
percent of cytotoxic T lymphocytes | 0.09 [0 to 0.15] | 0.02 [0 to 0.14]
Statistical Analysis 1: Comparison: GM-CSF vs NPS+GM-CSF; Test type: Superiority; p = 0.71, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Intra-tumoral Tumor-infiltrating Lymphocytes (iTILs) Within the Basement Membrane
Description: Change from baseline in the iTILs at surgical resection. Wilcoxon rank sum test exact P-value was used.
Time Frame: Baseline to surgical resection, up to 5 weeks
Measure: Median (Inter-Quartile Range); unit: percent of iTILs
Arm/Group | GM-CSF | NPS+GM-CSF
Number analyzed (Participants) | 3 | 5
percent of iTILs | 0 [-0.5 to 3.0] | 0.5 [-0.3 to 0.5]
Statistical Analysis 1: Comparison: GM-CSF vs NPS+GM-CSF; Test type: Superiority; p = 0.964, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: Intra-tumoral Tumor-infiltrating Lymphocytes (iTILs)
Description: Change from baseline in the iTILs at surgical resection. Wilcoxon rank sum test exact P-value was used.
Time Frame: Baseline to surgical resection, up to 5 weeks
Measure: Median (Inter-Quartile Range); unit: percent of iTILs
Arm/Group | GM-CSF | NPS+GM-CSF
Number analyzed (Participants) | 3 | 5
percent of iTILs | 0 [-5 to 0] | 0 [-17.5 to 14.5]
Statistical Analysis 1: Comparison: GM-CSF vs NPS+GM-CSF; Test type: Superiority; p = 1, Wilcoxon (Mann-Whitney)

4. Secondary Outcome: Number of Participants With HER2 Expression in Biopsy and Resection Specimens
Description: Difference in HER2 Expression in Biopsy and Resection Specimens. Differences were assessed using a Fisher's exact test.
Time Frame: Baseline to surgical resection, up to 5 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | GM-CSF | NPS+GM-CSF
Number analyzed (Participants) | 4 | 9
Participants
  HER2 expression - biopsy 1+ | 2 | 3
  HER2 expression - biopsy 2+ | 2 | 0
  HER2 expression - biopsy 3+ | 0 | 3
  HER2 expression - biopsy Normal Breast Tissue | 0 | 1
  HER2 expression - biopsy Missing | 0 | 3
  HER2 expression - resection 1+ | 2 | 1
  HER2 expression - resection 2+ | 1 | 1
  HER2 expression - resection 3+ | 1 | 2
  HER2 expression - resection Normal Breast Tissue | 0 | 3
  HER2 expression - resection Missing | 0 | 2
Statistical Analysis 1: Comparison: GM-CSF vs NPS+GM-CSF; Test type: Other; p = 0.172, Fisher Exact — HER2 expression - biopsy
Statistical Analysis 2: Comparison: GM-CSF vs NPS+GM-CSF; Test type: Other; p = 0.38, Fisher Exact — HER2 expression - resection

5. Secondary Outcome: Number of Adverse Events, Graded According to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version (v) 4.03
Description: The number of serious and non serious adverse events for both arms. Graded According to national Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version (v) 4.03.
Time Frame: 3-6 months after surgery
Measure: Number; unit: adverse events
Arm/Group | GM-CSF | NPS+GM-CSF
Number analyzed (Participants) | 4 | 9
adverse events
  Serious Adverse Events | 0 | 2
  Non Serious Adverse Events | 40 | 91

6. Secondary Outcome: Number of Participants With Presence of Ductal Carcinoma in Situ (DCIS)
Description: Presence of DCIS with Invasive Cancer.
Time Frame: At resection
Measure: Count of Participants; unit: Participants
Arm/Group | GM-CSF | NPS+GM-CSF
Number analyzed (Participants) | 4 | 9
Participants
  Not Present | 3 | 7
  Present | 1 | 2

7. Other Pre Specified Outcome: Immune Cell Analysis
Description: Will utilize tissue-based cyclic immunofluorescence (t-CyCIF), a novel, highly multiplexed imaging modality that follows the imaging of formalin-fixed, paraffin embedded (FFPE) tissue sections at subcellular resolution across 20-60 distinct antigen channels. 4-6 panels that will be used include both my not be limited to an already optimized immune panel.
Time Frame: up to 6 months after completion of the vaccination series timepoint
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Immune Infiltrates in Normal Tissue Maximally Distant From the Tumor (in Mastectomy Samples)
Description: In the mastectomy samples only will perform core needle biopsies of the normal tissue, maximally distant from the tumor (ex vivo after the mastectomy if performed and store for future studies of immune infiltrates.
Time Frame: Up to 6 months after completion of the vaccination series timepoint
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Toxicity Profile According to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version (v) 4.03)
Time Frame: up to 3 months after surgery
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Degree of Lymphocyte Infiltration
Description: We will define intra-tumoral TIL as those within the basement membrane. Stromal TIL will be defined as those in the periductal/lobular stroma including the intralobular stromal infiltrate. Cells in the interlobular stromal inflammatory infiltrate will be excluded. All mononuclear cells will be scored but polymorphonuclear leukocytes will be excluded. Intra-tumoral and stromal TILs will be scored as a continuous variable and the percentage of in the surgical specimen will be compared to that in the pre-vaccination diagnostic biopsy.
Time Frame: Up to 6 months after completion of the vaccination series timepoint
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: adverse events were assessed from randomization to the final follow up visit up to 8 months
Arm/Group | GM-CSF | NPS+GM-CSF
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/9
Serious Adverse Events (participants affected / at risk) | 2/4 | 0/9
Other Adverse Events (participants affected / at risk) | 4/4 | 9/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | GM-CSF (N=4) | NPS+GM-CSF (N=9)
Decreased Ejection Fraction (Cardiac disorders) | 1 | 0
Wound infection (Infections and infestations) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | GM-CSF (N=4) | NPS+GM-CSF (N=9)
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Allergic Reaction (Immune system disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 2
Breast Infection (Infections and infestations) | 0 | 1
Breast Pain (Reproductive system and breast disorders) | 2 | 3
Bruising (Injury, poisoning and procedural complications) | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Dermatitis radiation (Injury, poisoning and procedural complications) | 3 | 4
Erythema multiforme (General disorders) | 0 | 1
Fatigue (General disorders) | 0 | 2
Fever (General disorders) | 0 | 2
Flu like symptoms (General disorders) | 0 | 1
Headache (General disorders) | 1 | 1
Hot flashes (Vascular disorders) | 0 | 1
Hypertension (Vascular disorders) | 0 | 1
Injection Site reaction (General disorders) | 4 | 9
Musculoskeletal and connective tissue disorder- other (Musculoskeletal and connective tissue disorders) | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 2
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pain (General disorders) | 2 | 1
Pruritus (General disorders) | 3 | 3
Seroma (Surgical and medical procedures) | 0 | 1
Sinus Tachycardia (Cardiac disorders) | 0 | 1
Sinusitis (Infections and infestations) | 0 | 2
Mild Folliculitis (Skin and subcutaneous tissue disorders) | 0 | 1
Skin Hyperpigmentation (Skin and subcutaneous tissue disorders) | 2 | 3
Sore Throat (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Surgical and Medical Procedures Other (Surgical and medical procedures) | 0 | 2
Urinary Tract Infection (Infections and infestations) | 0 | 1
Vaginal Discharge (Reproductive system and breast disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-10-24): https://cdn.clinicaltrials.gov/large-docs/82/NCT02636582/Prot_SAP_000.pdf